CLINICAL TRIAL: NCT00140686
Title: A Multi-country & Multi-center Study to Assess the Efficacy, Safety & Immunogenicity of 2 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Infants in Co-administration With Specific Childhood Vaccines
Brief Title: To Test 2 Doses of GSK Biologicals' Oral Live Attenuated Human Rotavirus (HRV) Vaccine in Healthy Infants in Co-administration With Specific Childhood Vaccines
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 102247/036
Record Dates: First submitted 2005-08-31; First posted 2005-09-01 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Infections, Rotavirus
MeSH Terms: conditions — Rotavirus Infections | interventions — Rotavirus Vaccines

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

INTERVENTIONS:
Biological: Rotavirus (vaccine)

SUMMARY:
The main objectives of this study is to determine vaccine efficacy against any rotavirus (RV) gastroenteritis (GE) during the first efficacy period.

DETAILED DESCRIPTION:
The study has two groups: Group HRV and Group Placebo. Two oral doses administered to healthy infants who are 6-14 weeks of age at the time of Dose 1, according to a 0, 1 to 2-month schedule. Routine EPI vaccinations are given at the discretion of the investigator and according to local National Plans of Immunisation schedule in each participating country.

ELIGIBILITY:
Inclusion criteria:

* Healthy infants 6 -14 weeks of age at the time of the first study vaccination with birth weight > 2000g whose parent/guardian sign a written informed consent and whose parents/guardians can and will comply with the requirements of the protocol (e.g., completion of the diary cards, return for follow-up visits).

Exclusion criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration of a vaccine not foreseen by the study protocol within 14 days before each dose of study vaccine(s) and ending 14 days after.
* Chronic administration (defined as more than 14 days) of immunosuppressants since birth. (Topical steroids are allowed.)
* History of diphtheria, tetanus, pertussis, Hib disease and/ or hepatitis B disease (in all subjects). Only for subjects in Spain: history of meningococcal group C disease. Only for subjects in France and Germany: history of disease caused by Streptococcus pneumoniae.
* History of use of experimental rotavirus vaccine.
* Previous vaccination against diphtheria, tetanus, pertussis, Haemophilus influenzae type b (in all subjects). Only for subjects in Spain: previous vaccination against meningococcal group C. Only for subjects in France and Germany: previous vaccination against Streptococcus pneumoniae.
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the GI tract, IS or other medical condition determined to be serious by the investigator.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination (no laboratory testing is required).
* History of allergic disease or reaction likely to be exacerbated by any component of the vaccine.
* Acute disease at the time of enrolment. (Acute disease is defined as the presence of a moderate or severe illness with or without fever. All vaccines can be administered to persons with a minor illness such as mild upper respiratory infection with or without low-grade febrile illness, i.e. Oral temperature <37.5°C (99.5°F) / Axillary temperature <37.5°C (99.5°F) / Rectal temperature <38°C (100.4°F).)
* Gastroenteritis within 7 days preceding the first study vaccine administration (warrants deferral of the vaccination).
* A family history of congenital or hereditary immunodeficiency.
* Administration of immunoglobulins and/or blood products since birth or planned administration during the study period.
* History of any neurologic disorders or seizures.
* Acute or chronic, clinically significant pulmonary, cardiovascular, hepatic or renal functional abnormality, as determined by physical examination or laboratory screening tests.

Ages: 6 Weeks to 14 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 3994 (Actual)
Dates: Start 2004-09; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

PRIMARY OUTCOMES:
Occurrence of any RV GE caused by the circulating wild-type RV strains during the first efficacy follow-up period.

SECONDARY OUTCOMES:
Occurrence of severe RV GE caused by the circulating wild-type RV strains during the each efficacy follow-up period.
Occurrence of any and severe RV GE caused by the circulating wild-type RV strains of G1 serotype during each efficacy follow-up period.
Occurrence of any and severe RV GE caused by the circulating wild-type RV strains of non-G1 serotypes during each efficacy follow-up period.
Occurrence of hospitalization due to RV GE caused by the circulating wild-type RV strains during each efficacy follow-up period.
Occurrence of any medical attention (medical provider contact, advice, visit; emergency room contact or visit or hospitalization) for RV GE caused by the circulating wild-type RV strains during each efficacy follow-up period.
Occurrence of any and severe RV GE caused by the circulating wild-type RV strains during the period starting from Dose 1 of the study vaccine until Visit 5.
Occurrence of any and severe RV GE caused by the circulating wild-type RV strains during the first efficacy follow-up period in subjects who completed the two-dose vaccination course before the RV epidemic season.
Occurrence of any and severe RV GE caused by the circulating wild-type RV strains during the first efficacy follow-up period in subjects who were vaccinated during the RV epidemic season.
Immune response to HRV vaccine at Visit 1 and Visit 3.
Immune response to all antigens contained in each of the different childhood vaccines at Visit 3 and Visit 4 or Visit 6 (if applicable):
In a subset of subjects (N=1800), occurrence of each type of solicited symptom within the 8-day solicited follow-up period (Day 0 to Day 7) after each dose of HRV/placebo.
For all subjects, occurrence of unsolicited symptoms within 31 days (Day 0 to Day 30) after each dose of HRV/placebo and SAEs throughout the entire study period.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (94):
- Czechia (10):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Havlíčkův Brod
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Humpolec
  - GSK Investigational Site, Jindřichův Hradec
  - GSK Investigational Site, Náchod
  - GSK Investigational Site, Ostrava
  - GSK Investigational Site, Pardubice
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Znojmo
- Finland (16):
  - GSK Investigational Site, Espoo
  - GSK Investigational Site, Helsinki
  - GSK Investigational Site, Hyvinkää
  - GSK Investigational Site, Jarvenpaa
  - GSK Investigational Site, Jyväskylä
  - GSK Investigational Site, Kokkola
  - GSK Investigational Site, Kotka
  - GSK Investigational Site, Kuopio
  - GSK Investigational Site, Lahti
  - GSK Investigational Site, Oulu
  - GSK Investigational Site, Pori
  - GSK Investigational Site, Riihimäki
  - GSK Investigational Site, Seinäjoki
  - GSK Investigational Site, Tampere
  - GSK Investigational Site, Turku
  - GSK Investigational Site, Vantaa
- France (20):
  - GSK Investigational Site, Boulogne
  - GSK Investigational Site, Chambéry
  - GSK Investigational Site, Châlons-en-Champagne
  - GSK Investigational Site, Courbevoie
  - GSK Investigational Site, Draguignan
  - GSK Investigational Site, Essey-lès-Nancy
  - GSK Investigational Site, Floirac
  - GSK Investigational Site, Gradignan
  - GSK Investigational Site, Issy-les-Moulineaux
  - GSK Investigational Site, Le Havre
  - GSK Investigational Site, Les Lilas
  - GSK Investigational Site, Manosque
  - GSK Investigational Site, Maromme
  - GSK Investigational Site, Maurepas
  - GSK Investigational Site, Nogent-sur-Marne
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rosny-sous-Bois
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Saint-Quentin
  - GSK Investigational Site, Thionville
- Germany (30):
  - GSK Investigational Site, Birkenfeld, Baden-Wurttemberg
  - GSK Investigational Site, Mannheim, Baden-Wurttemberg
  - GSK Investigational Site, Oberkirch, Baden-Wurttemberg
  - GSK Investigational Site, Freising, Bavaria
  - GSK Investigational Site, Kaufering, Bavaria
  - GSK Investigational Site, Munich, Bavaria
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Eschwege, Hesse
  - GSK Investigational Site, Fulda, Hesse
  - GSK Investigational Site, Wiesbaden, Hesse
  - GSK Investigational Site, Salzgitter, Lower Saxony
  - GSK Investigational Site, Wolfenbüttel, Lower Saxony
  - GSK Investigational Site, Bützow, Mecklenburg-Vorpommern
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Detmold, North Rhine-Westphalia
  - GSK Investigational Site, Espelkamp, North Rhine-Westphalia
  - GSK Investigational Site, Goch, North Rhine-Westphalia
  - GSK Investigational Site, Gütersloh, North Rhine-Westphalia
  - GSK Investigational Site, Löhne, North Rhine-Westphalia
  - GSK Investigational Site, Minden, North Rhine-Westphalia
  - GSK Investigational Site, Oberhausen, North Rhine-Westphalia
  - GSK Investigational Site, Velbert, North Rhine-Westphalia
  - GSK Investigational Site, Willich, North Rhine-Westphalia
  - GSK Investigational Site, Trier, Rhineland-Palatinate
  - GSK Investigational Site, Cossebaude, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Flensburg, Schleswig-Holstein
  - GSK Investigational Site, Glücksburg, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (4):
  - GSK Investigational Site, Bari, Apulia
  - GSK Investigational Site, Rome, Lazio
  - GSK Investigational Site, Genoa, Liguria
  - GSK Investigational Site, Ragusa, Sicily
- Spain (14):
  - GSK Investigational Site, Almería
  - GSK Investigational Site, Baracaldo (Vizcaya)
  - GSK Investigational Site, Barakaldo
  - GSK Investigational Site, Barcelona
  - GSK Investigational Site, Berango (Vizcaya)
  - GSK Investigational Site, Bilbao
  - GSK Investigational Site, Blanes
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Móstoles/Madrid
  - GSK Investigational Site, Munguía (Vizcaya)
  - GSK Investigational Site, San Vicent Dels Horts
  - GSK Investigational Site, Sant Adriá de Beyós, Barcelona
  - GSK Investigational Site, Sant Eugenia de Berga, Barcelona
  - GSK Investigational Site, Sodupe (Vizcaya)

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] De Vos B, Han HH, Bouckenooghe A, Debrus S, Gillard P, Ward R, Cheuvart B. Live attenuated human rotavirus vaccine, RIX4414, provides clinical protection in infants against rotavirus strains with and without shared G and P genotypes: integrated analysis of randomized controlled trials. Pediatr Infect Dis J. 2009 Apr;28(4):261-6. doi: 10.1097/INF.0b013e3181907177. PMID 19289978
- [Background] Soriano-Gabarró M et al. (2008) Potential impact of Rotarix according to rotavirus type distribution. Pediatr Infect Dis J. 27(1) Supplement: S28-S32.
- [Background] Vesikari T, Karvonen A, Prymula R, Schuster V, Tejedor JC, Cohen R, Meurice F, Han HH, Damaso S, Bouckenooghe A. Efficacy of human rotavirus vaccine against rotavirus gastroenteritis during the first 2 years of life in European infants: randomised, double-blind controlled study. Lancet. 2007 Nov 24;370(9601):1757-63. doi: 10.1016/S0140-6736(07)61744-9. PMID 18037080
- [Background] Vesikari T, Prymula R, Schuster V, Tejedor JC, Cohen R, Bouckenooghe A, Damaso S, Han HH. Efficacy and immunogenicity of live-attenuated human rotavirus vaccine in breast-fed and formula-fed European infants. Pediatr Infect Dis J. 2012 May;31(5):509-13. doi: 10.1097/INF.0b013e3182489cac. PMID 22228235
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Annotated Case Report Form: 102247/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 102247/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 102247/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 102247/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 102247/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 102247/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 102247/036 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register